CLINICAL TRIAL: NCT05204082
Title: Use of SU-VEID™ As An Adjunct to Vein Visualization Technology to Improve Peripheral Venous Access Success in Children
Brief Title: A Study to Evaluate SU-VEID™ for Improving Peripheral Venous Access Success in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The available SU-VEID devices expired and unable to acquire additional devices for study completion.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael E. Nemergut, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-006822
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Intravenous Access

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard IV Insertion (No Intervention): Pediatric patients in surgical pre-op requiring an IV catheter for surgery will have standard IV insertion
- SU-VEID assisted IV Insertion (Other): Pediatric patients in surgical pre-op requiring an IV catheter for surgery will have IV insertion using SU-VEID device
  Interventions: Device: Single Use Vein Entry Indicator Device

INTERVENTIONS:
Device: Single Use Vein Entry Indicator Device — Electronic pressure sensing device, integrated to a conventional needle catheter, and which indicates continuously during intravenous cannulation whether the tip of the needle is inside or outside of a vein, to assist a clinician in intravenous cannulation.
  Other Names: SU-VEID
  Arms: SU-VEID assisted IV Insertion

SUMMARY:
The purpose of this study is to determine if use of the SU-VEID™ in children facilitates an increase success rate of peripheral intravenous starts, in comparison to the conventional method of vein entry techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patient age < 18 years old.
* Pediatric patients in surgical pre-op (0-18 years old), requiring an I.V. catheter for surgery who are difficult venous access.
* Written informed consent/ assent from the patient or legal guardian.

Exclusion Criteria:

- Patient age > 18 years old.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 169 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Nemergut, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard IV Insertion | SU-VEID Assisted IV Insertion
Started | 84 | 85
Completed | 84 | 85
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard IV Insertion | SU-VEID Assisted IV Insertion | Total
Number analyzed (Participants) | 84 | 85 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.31 (3.99) | 5.35 (4.19) | 5.33 (4.086)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 48 | 49 | 97
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 84 | 85 | 169

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With IV Access at First Attempt
Description: Percentage of participants to have an IV access within the first attempt when using the SU-VEID Device in comparison to the conventional procedure
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Standard IV Insertion | SU-VEID Assisted IV Insertion
Number analyzed (Participants) | 84 | 85
percentage of participants | 70.2 | 67.1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 1 day on all participants.
Arm/Group | Standard IV Insertion | SU-VEID Assisted IV Insertion
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/85
Other Adverse Events (participants affected / at risk) | 0/84 | 0/85

LIMITATIONS AND CAVEATS:
Study terminated due to the the available SU-VEID devices expiring and the inability to acquire additional devices for study completion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT05204082/Prot_SAP_000.pdf